Official Title: Effects of a Rheumatoid Arthritis Self-management program-a Randomized

**Controlled Trial** 

NCT number: NCT03470740 Date of the document: 20160801

## **Background**

Rheumatoid arthritis (RA) is a persistent systemic disease (Flurey et al., 2014; WHO, 2003). The prevalence of RA is 0.3% - 1% worldwide (WHO, 2003), and 0.6% in Taiwan (Chou, 2003). Within a decade of its onset, RA leads to work disability defined as a total cessation of employment in between 51% and 59% of patients (WHO, 2003). In Taiwan, the Ministry of Health and Welfare (2014) emphasized that people suffer from knee joint degeneration is up to 15% prevalence, and the most common cause including RA. WHO (2003) commented that although the mortality rate of RA is low, a decreased life expectancy is associated with some musculoskeletal disorders, inflammation of the multi-system, and ischemic heart disease. The impact of RA including reduction of patients' daily activities, effects on the different dimensions of the quality of life, reduce work capacity (Lee et al., 2010; WHO, 2003), and significant increase health care costs (Furner et al., 2011). Epidemiological data indicate that individuals with RA are most often diagnosed in their 40s (Lin et al., 2004). With the disease continuing into old age, we can anticipate that the number of older patients with RA is increasing on a worldwide basis. In Taiwan, the life expectancy is increase and the average life span achieves 79.84-year (Ministry of the Interior, 2015), and indicate that individuals with RA need to live with the disease for more than 40 years.

Patients' involvement in the management of their care is referred to as self-management, which has been defined by Barlow and colleagues (2002, p.178) as "the individual's ability to manage the symptoms, treatment, physical and psychosocial consequences and life style changes inherent in living with a chronic condition". Barlow further states that for SM to be effective, it needs to encompass the ability to monitor one's condition and to affect the behavioral and emotional responses necessary to maintain a satisfactory quality of life. This definition implies that SM is more than simple adherence to treatment guidelines because it incorporates the psychological and social management of living with a chronic illness. SM involves, on the patient's part, acquiring the knowledge, practicing the skills and developing the confidence to deal with disease-related problems, and making and maintaining behavioral changes to maximize well-being (Dures & Hewlett, 2012). Chronic diseases such as RA and related conditions have no 'cure', the goal of intervention is to minimize disease impact and optimize physical, emotional, and social health (Keysor et al., 2001). Day-to-day SM is extremely important in achieving optimal health outcomes, and people with arthritis use a variety of strategies to relieve symptoms or manage disease consequences (Keysor et al., 2001). Hence, SM in arthritis tends to adopt a more holistic approach including management of psychosocial consequences and life style changes (Barlow et al., 2002).

#### **Methods**

### Research Design

An *experimental design* was used to examine the effectiveness of a SM intervention for RA patients.

## Sample and Setting

A medical center in northern Taiwan was selected as the research setting to ensure sufficient numbers of RA patients are able to be recruited for this study, and the teaching hospital is constantly striving to improve their services, and is readily accessible to the researcher. Patients who visited the rheumatology departments of the medical center was eligible for the study and the inclusion criteria include: (1) diagnosed with RA, (2) age of 20 years or over, (3) disease considered by the treating rheumatologist to have been stable for at least 3 months, and (4) able to understand and comply with the study treatment. Patients were excluded if they are suffering from other terminal illnesses, severe dementia or another debilitating psychiatric disorder, living in a long-term care facility, and participation in another research protocol. All patients were under the medical care of their rheumatologist during the study.

# Sampling Procedure

Patients were approached for recruitment when they visit in the medical center rheumatology departments. If the patients meet the inclusion criteria and agree to participate in the study then randomly assigned to the experimental and control groups were proceeded using a computerized allocation procedure in SPSS 17.0 for Windows by an independent researcher. A numbered envelope was given. The big and opaque envelopes were numbered from 1 to 260 and contained the baseline data collection questionnaires and another sealed of small opaque envelope. The small opaque envelope contained a randomly determined using the computer-generated sequence of random numbers: number zero is for the control group and number one is for the experimental group. The researcher opened the big envelop and collect the baseline data, and then open the small sealed envelope to randomly assign participants to two groups. If the patient is random assigned to the control group, the usual care of the RA was received. Another experimental group received the program. For this sampling procedure, neither the researcher nor the participant is aware of treatment group assignment until after the baseline questionnaire has been collected. The CONSORT (Consolidated Standards of Reporting Trials) flow diagram (Moher et al., 2001) will be followed to manage the random allocation.

# Intervention Program

The intervention program was based on self-efficacy theory (Bandura, 1977, 1986, 2004), and the four resources of self-efficacy such as mastery experience, social modeling, social persuasion, and physical and emotional states will be incorporate to emphasize patients' knowledge, skill, and responsibility in managing their RA situations. Various sources of information affect efficacy judgments and influence how people weigh and integrate them into actions.

### Instruments and Outcome Measurements

Many of the standard measuring instruments selected have been used in previous studies of people with arthritis, and have established reliability and validity. Outcome data were collected at the baseline, and 2, 3, and 6 months including RA disease activity (DAS-28), arthritis self-efficacy (ASE), physical functioning (MHAQ), quality of life (SF-36), self-management behaviors, and and health care utilization.

#### Procedure and Data Collection

The researcher contacted the RA patients if they meet the inclusion criteria, and a face-to-face interview started. The researcher explained the purpose and procedure of the project, as well as the participants' rights and the benefits of participating. Next, participants agreeing to participate signed consent forms. Regarding collection the data, the baseline data was collected including background information, disease activity, arthritis self-efficacy, quality of life, physical functioning, self-management behaviors, and health care utilization. It followed questionnaire guide to collect data, and the person who collected the data and the researcher who visit the patient for the intervention was never the same. After completion of baseline data, patients were randomly allocated to the intervention or control group by an independent researcher. Control patients received usual care, and the intervention group received the 6-week RA self-management program. All participants were followed up for 6 months, and the data were all collected at the RA OPD when patients were back to the clinic.

# Data Analysis

Data were double entered for verification and the level of significance was set at alpha of .05 using SPSS Version 17.0. Descriptive statistical analyses were used to establish baseline characteristics of RA patients using means, ranges, standard deviations, frequencies, and percentages. Background characteristics and outcomes at baseline were compared between two groups by means of chi-square tests and t-tests for independent samples. To evaluate the effect of the intervention over the total follow-up period, we used the multiple linear regression method used in the *GEE* (Liang & Zeger, 1986) to take into account of internal dependencies within subjects (due to the repeated measurements) and to adjust for the effects of certain factors. Effects evaluated included the main effects of time and group and two-way interaction effect(s) of time by group. A significant interaction effect of time by group would indicate a significant change from baseline to a specific later time point between the two groups. Significant interaction effect(s) in GEE results would provide evidence of intervention effects.

## **Ethical Considerations**

The study was reviewed and approved by the Institutional Review Boards of the hospitals of the PI prior to data collection. The participants were informed both orally and in writing about the purpose of the study, assured that participation was voluntary, and the benefits of participating. To ensure the security of the intervention, the researcher discussed with the physician about the potential participants' condition and their self-management. They signed the informed consent, was guaranteed confidentiality, and was assured an anonymous presentation of the findings.

#### References

- Albanoa, M.G., Giraudet-Le Quintrec, J. S., Crozet, C., & d'Ivernois, J. F. (2010). Characteristics and development of therapeutic patient education in rheumatoid. *Joint Bone Spine*, 77, 405-410.
- Bandura, A. (1977). Social learning theory. Englewood Cliffs, NJ: Prentice Hall.
- Bandura, A. (1997). Self-efficacy: the exercise of control. New York: Freeman.
- Bandura, A. (2004). Swimming against the mainstream: the early years from chilly tributary to transformative mainstream. *Behaviour Research and Therapy, 42*(6), 613-630.
- Barlow J, Wright C, Sheasby J, Turner A, Hainsworth J. (2002). Self-management approaches for people with chronic conditions: a review. *Patient Education and Counselling*, 48, 177-187.
- Barlow, J.H., Williams, B., & Wright, C. C. (1997a). Improving arthritis self-management among older adults: 'Just what the doctor didn't order'. *British Journal of Health Psychology*, **2**, 175–186.
- Barlow, J. H., Williams, B., & Wright, C. C. (1997b). The reliability and validity of the arthritis self-efficacy scale in a UK context. *Psychology Health and Medicine*, *2*(1), 3-17.
- Breedland, I., van Scheppingen, C., Leijsma, M., Verheij-Jansen, N. P., & van Weert, E. (2011). Effects of a group-based exercise and educational program on physical performance and disease self-management in rheumatoid arthritis: a randomized controlled study. *Physical Therapy*, 91,879-893.
- Burckhardt, C. S. (2005). Educating patients; Self-management approaches. *Disability and Rehabilitation*, 27(12), 703-709.
- Burke, L. E., Dunbar-Jacob, J. M., & Hill, M. N. (1997). Compliance with cardiovascular disease prevention strategies: a review of the research. Ann Behav Med, *19*(3), 239-263.
- Chou CD (ed.) (2003) Rheumatology. CO-CHI, Taipei.
- Conn, D. L., Pan, Y., Easley, K. A., Comeau, D. L., Carlone, J. P., Culler, S. D., & Tiliakos, A. (2013). The effect of the Arthritis Self-Management Program on outcome in African Americans with rheumatoid arthritis served by a public hospital. *Clin Rheumatol*, 32, 49-59.
- Dougados, M., Soubrier, M., Perrodeau, E., Gossec, L., Fayet, F., Gilson, M.,...Ravaud, P. (2015). Impact of a nurse-led programme on comorbidity management and impact of a patient selfassessment of disease activity on the management of rheumatoid arthritis. Annals of the Rheumatic Diseases, 74, 1725-1733.
- Dures, E., & Hewlett, S. (2012). Cognitive-behavioural approaches to self-management in rheumatic disease, *Nature Reviews Rheumatology*, 8, 553-559.
- Flurey, C. A., Morris, M., Richards, P., Hughes, R., & Hewlett, S. (2014). It's like a juggling act: rheumatoid arthritis patient perspectives on daily life and flare while on current treatment regimes. *Rheumatology*, *53*, 696-703.
- Furner, S. E., Hootman, J. M., Helmick, C. G., Bolen, J., & Zack, M. M. (2011). Health-related quality of life of U.S. Adults with arthritis: analysis of data from the behavioral risk factor surveillance system, 2005, and 2007. *Arthritis Care Res* 2003, 2011, 788-799.

- Hammond, A., Bryan, J. & Hardy, A. (2008). Effects of a modular behavioural arthritis education programme: a pragmatic parallel-group randomized controlled trial. *Rheumatology (Oxford)* 47, 1712-1718.
- Hampson, S. E., Glasgon, R. E., Zeiss, A.M., Birskovich, S. F., Foster, L., & Lines, A. (1993). Self-management of osteoarthritis. *Arthritis Care and Research*, 6, 17 22.
- Hewlett, S., Ambler, N., Almeida, C., Cliss, A., Hammond, A., Kitchen, K., ...Pollock, J. (2011). Self-management of fatigue in rheumatoid arthritis: a randomised controlled trial of group cognitive-behavioural therapy. *Ann. Rheum. Dis.* 70, 1060–1067.
- Kett, S., Flint, J., Openshaw, M., Raza, K., & Kumar, K. (2010). Self-management strategies used during flares of rheumatoid arthritis in an ethnically diverse population. *Musculoskelet. Care*, 8, 204-214.
- Keysor, J. J., Currey, S. S., & Callahan, L. F. (2001). Behavioral aspects of arthritis and rheumatic disease self-management. *Dis Manage Health Outcomes*, 9(2), 89-98.
- Köse, S. K., Ö ztuna D., Kutlay, S., Elhan, A. H., Tennant, A., & Küçükdeveci, A. A. (2010). Psychometric properties of the HealthAssessment Questionnaire Disability Index (HAQ-DI) and the Modified Health AssessmentQuestionnaire (MHAQ) in patients with knee osteoarthritis. *Turkish Journal of Rheumatology*, 25(3), 147-155.
- Lee, H-C., Tsai, Y-F., Luo, S-F., & Tsay, P-K. (2010). Predictors of disability in Taiwanese patients with rheumatoid arthritis, *Journal of Clinical Nursing*, 19, 2989-2996.
- Liang, K. Y., & Zeger, S. L. (1986). Longitudinal data analysis using generalized linear models. *Biometrika*, 73(1), 13-22.
- Lin, Y. C., Liao, H. T., Liang, T. H., & Lin, H. Y. (2004). The pitfalls in the diagnosis and treatment of rheumatic disease. *Journal of Internal Medicine of Taiwan*, 15(4), 147–160.
- Liu Y.-J., Xu H.-P., & Zhao H. (2011). Self-management approaches following total knee arthroplasty. *Journal of Clinical Rehabilitative Tissue Engineering Research*, *15*(17), 3057-3061.
- Liu, G., & Liang, K. Y. (1997). Sample size calculations for studies with correlated observations. *Biometrics*, *53*(3), 937-947.
- Lorig, K., & Laurent, D. (2007). Stanford Patient Education Research Center (2007). Primer for evaluating outcomes. Retrieved Nov. 9, 2012, from <a href="http://patienteducation.stanford.edu/research/primer.html">http://patienteducation.stanford.edu/research/primer.html</a>
- Lorig, K., Chastain, R. L., Ung, E., Shoor, S., & Holman, H. R. (1989a). Development and evaluation of a scale to measure self-efficacy in people with arthritis. *Arthritis and Rheumatism*, 32(1), 37-44.
- Lorig, K., Seleznick, M., Lubeck, D., Ung, E., Chastain, R., & Holman, H. (1989b). The beneficial outcomes of the arthritis self-management course are not adequately explained by behavior change. *Arthritis Rheum*, 32, 91-95.
- Lorig, K.R., Sobel, D.S., Ritter, P.L., Laurent, D., & Hobbs, M. (2001). Effect of a self-management

- program on patients with chronic disease. Effective Clinical Practice, 4, 256-262.
- Lu, J. F. R., Lan, C. F., Wu, S. C., Liu, W. L., Lee, J. L., & Chi, C. H. (1996). SF-36, From http://sf36.cgu.edu.tw/. (accessed December, 2011).
- Lu, S-R., Lin, H-Y., Lin, K-C., & Lin, H. R. (2008). Quality of life in middle-aged and older Taiwanese patients with rheumatoid arthritis. *Journal of Nursing Research*, 16(2), 121-130.
- Lynn, M. (1986). Determination and quantification of content validity. *Nursing Research*, 35, 382-385.
- McDowell, J., Courtney, M., Edwards, H. & Shortridge-Baggett, L. (2004). International collaboration in promoting self-management of chronic disease, in Dept of Health and Ageing (ed) *National Chronic Condition Self-Management Conference Proceedings*. pp. 368 -371. Commonwealth of Australia: Canberra.
- Ministry of Health and Welfare (2014). Health and Welfare Ministry focus news. Retrieved from http://www.mohw.gov.tw/cht/Ministry/RSSDetail.aspx?op=news on 1 December 2014.
- Ministry of the Interior. (2015). latest statistics. Retrieved from http://www.moi.gov.tw/stat/chart.aspx on 1 December 2015.
- Moher, D., Schulz, K. F., & Altman, D. G. (2001). The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. *BMC Medical Research Methodology*, *1*(2), 1-7.
- Newman, S., Steed, L., & Mulligan, K. (2004). Self-management interventions for chronic illness. *Lancet*, *364*, 1523-1537.
- Parlar, S., Fadiloglu, C., Argon, G., Tokem, Y., & Keser, G. (2013). The effects of self-pain management on the intensity of pain and pain management methods in arthritic patients. *Pain Management Nursing*, *14* (3), 133-142.
- Prevoo, M. L., van't Hof, M. A., Kuper, H. H., van Leeuwen, M. A., van de Putte, L. B., van Riel, P. L. (1995). Modified disease activity scores that include twenty-eight-joint counts Development and validation in a prospective longitudinal study of patients with rheumatoid arthritis. *Arthritis and Rheumatism*, 38(1), 44-48.
- Ritter, P.L., Kaymaz, H., Stewart, A., Sobel, D.S., Lorig, K.R. (2001). Self-reports of health care utilization compared to provider records. *Journal of Clinical Epidemiology*, *54*, 136-141.
- Rosal, M. C., Ayers, D., Li, W., Oatis, C., Borg, A., Zheng, H., & Franklin, p. (2011). "A Randomized Clinical Trial of a Peri-Operative Behavioral Intervention to Improve Physical Activity Adherence and Functional Outcomes following Total Knee Replacement. *BMC Musculoskeletal Disorders*, 12(226), 1-7.
- Salaffi,F.,Cimmino,MA.,Leardini,G.,Gasparini,S.,&Grassi,W.(2009).Disease activity assessment of rheumatoid arthritis in daily practice: validity, internal consistency, reliability and congruency of the Disease Activity Score including 28 joints (DAS28) compared with the Clinical Disease Activity Index (CDAI). *Clinical and Experimental Rheumatology*, 27, 552-559.
- Scott, D. L., & Steer, S. (2007). The course of established rheumatoid arthritis. Best Pract Res Clin

- Rheumatol, 21, 943 -967.
- Shao, J. H., Chang, A. M., Edwards, H., Shyu, Y. I. L., & Chen, S. H. (2013). A randomized controlled trial of self-management programme improves health-related outcomes of older people with heart failure. *Journal of Advanced Nursing*, 69(11), 2458–2469.
- Shyu, Y. I. L., Lu, J. F. R., & Chen, S. T. (2009). Psychometric testing of the SF-36 Taiwan version on older stroke patients. *Journal of Clinical Nursing*, *18*(10), 1451-1459.
- Stanford Chronic Disease Self-Management Study (1996). Psychometrics reported in: Lorig K, Stewart A,Ritter P,González V,Laurent D,& Lynch J, *Outcome Measures for Health Education and other Health Care Interventions*. Thousand Oaks CA: Sage Publications, 24-25.
- Tsay, S. L. (2003). Self-efficacy training for patients with end-stage renal disease. *Journal of Advanced Nursing*, 43(4), 370-371.
- van den Akker-Scheek, I., Stevens, M., Groothoff, J. W., Bulstra, S. K., & Zijlstra, W. (2007). Preoperative or postoperative self-efficacy: Which is a better predictor of outcome after total hip or knee arthroplasty? *Patient Education and Counseling*, 66(1), 92-99.
- van der Heijde, D. M., van't Hof, M. A., van Riel, P. L., Theunisse, L. A., Lubberts, E. W., van Leeuwen, M. A., ... van de Putte, L. B. (1990). Judging disease activity in clinical practice in rheumatoid arthritis: first step in the development of a disease activity score. *Annals of the Rheumatic Disease*, 49(11), 916-920.
- van Gestel, A. M., Haagsma, C. J., & van Riel, P. L. (1998). Validation of rheumatoid arthritis improvement criteria that include simplified joint counts. *Arthritis Rheum*, 41(10),1845-1850.
- Ware, J. E. Jr., & Sherbourne, C. D. (1992). The MOS 36-item short-form health survey (SF-36). Conceptual framework and item selection, *Med Care*, 30, 473-483.
- Ware, J. E. Jr., (2011). SF-36 Health Survey, From Update http://www.sf-36.org/tools/SF36.shtml#MODEL.
- Williams, K. E., & Bond, M. J. (2002). The roles of self-efficacy, outcome expectancies and social support in the self-care behaviours of diabetics. *Psychology Health & Medicine*, 7, 127-141.
- World Health Organization. (2003). The Burden of Musculoskeletal Conditions at the Start of the New Millennium. Available at: http://whqlibdoc.who.int/trs/WHO TRS 919.pdf
- Wu, S-F.V., Kao, M. J., Wu, M. P., Tsai, M. W., & Chang, W. W. (2011). Effects of an osteoarthritis self-management programme. *Journal of Advanced Nursing*, 67(7), 1491-1501.